CLINICAL TRIAL: NCT00570089
Title: Microvascular Coronary Disease In Women: Impact Of Ranolazine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: CV Therapeutics (Industry)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 10465
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Myocardial Ischemia
Keywords: Ranolazine; Myocardial ischemia; Double blinded; Placebo controlled
MeSH Terms: conditions — Myocardial Ischemia | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Drug Ranexa, Then Placebo (Experimental): Participants first received study drug Ranexa, 500mg, orally twice daily for 2 weeks, assuming tolerance, followed by 1000mg orally twice daily for an additional 2 weeks. If the participant is unable to increase dose secondary to side effects, she will remain on 500mg twice daily for the second 2-week interval.
  After a washout period of 2 weeks, they then received Placebo tablet (matching Ranexa tablet).
  Interventions: Drug: Ranolazine; Drug: Placebo
- Placebo, Then Study Drug Ranexa(Ranolazine) (Experimental): Participants first received Placebo tablet (matching Ranexa tablet) for two weeks.
  After washout period of 2 weeks, they then received Ranexa 500mg, orally twice daily for 2 weeks, assuming tolerance, followed by 1000mg orally twice daily for an additional 2 weeks. If the participant is unable to increase dose secondary to side effects, she will remain on 500mg twice daily for the second 2-week interval.
  Interventions: Drug: Ranolazine; Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — 500mg, orally twice daily for 2 weeks, assuming tolerance, followed by 1000mg orally twice daily for an additional 2 weeks. If the participant is unable to increase dose secondary to side effects, she will remain on 500mg twice daily for the second 2-week interval.
  Other Names: Ranexa
Drug: Placebo — Placebo, 500mg, orally twice daily for 2 weeks, assuming tolerance, followed by 1000mg orally twice daily for an additional 2 weeks. If the participant is unable to increase dose secondary to side effects, she will remain on 500mg twice daily for the second 2-week interval.

SUMMARY:
1. To evaluate the impact of ranolazine extended-release tablets in women with subendocardial ischemia due to microvascular endothelial dysfunction on myocardial ischemia (Cardiac Magnetic Resonance (CMR) extent, severity.
2. To evaluate the impact of ranolazine extended-release tablets in women with subendocardial ischemia due to microvascular endothelial dysfunction on the outcomes of angina (Seattle Angina Questionnaire (SAQ), WISE angina frequency, Duke Activity Status Inventory(DASI) and SF-36).

DETAILED DESCRIPTION:
Interested women will be considered for the study if they meet inclusion and exclusion criteria including review of baseline CMR, ECG and blood work (liver and kidney function). The baseline CMR must be completed within 12 months previous to enrollment.

Eligible women with angina and CMR subendocardial perfusion abnormalities, defined as CMR qualitative perfusion abnormalities of greater than or equal to 10% reported as abnormal following blind review per protocol, will be consented and enrolled. The women will complete baseline demographic and health history questionnaires, including the SAQ, Women's Ischemic Syndrome Evaluation (WISE) angina frequency, DASI and SF-36.

This study is a double-blind, placebo controlled, cross-over design in which treatment order to ranolazine and placebo will be randomly assigned. Note: The participant's usual medication regimen will be continued throughout study participation. Following enrollment into the study, participants will be randomized to treatment #1 (either placebo or ranolazine). Ranolazine will be dosed as 500 mg orally twice daily for 2 weeks and, assuming tolerance, followed by 1000 mg orally twice daily for an additional 2 weeks. If the participant is unable to increase dose secondary to side effects, she will remain on 500 mg twice daily for the second 2 week interval. The first end of treatment CMR (CMR 1) will be scheduled at the end of the 4th week of treatment, approximately 4 hours after the morning dose of study drug. At this visit (Vis 2), concurrent medications, symptoms, and adverse events will be reviewed. Clinical measurements will be taken (weight, BP, waist and hip circumference) and questionnaires will be completed (SAQ, WISE angina frequency, DASI and SF-36).

After the first course of study treatment, the patient will undergo a two week wash-out with no study drug while continuing usual medication regimen. Following the washout period, study participants will start the second cycle of study drug treatment (i.e., the other study drug not received in treatment 1). At visit 3, participants will undergo baseline 2 measurements which include concurrent medication and symptom assessment, clinical measurements (weight, BP, waist and hip circumference) and will complete baseline 2 questionnaires (SAQ, WISE angina frequency, DASI and SF-36). Study drug treatment #2 will follow the same escalation of study drug dose as described above for treatment 1. The final study CMR (CMR 2) will be scheduled at the end of the 4th week of treatment 2, approximately 4 hours after the morning dose of study drug. At this visit (Vis 4), concurrent medications, symptoms, and adverse events will be reviewed. Clinical measurements will be taken (weight, blood pressure, waist and hip circumference) and questionnaires will be completed (SAQ, WISE angina frequency, DASI and SF-36). [See Table 1 for a listing of all study procedures by visit.] The two post study drug treatment CMRs will be performed at the same time of day, replicating temperature, fasting state, adenosine dosing and infusion, magnet settings and using the same over-reader. The dose of adenosine will be consistent for all study CMR tests: 140 mcg/kg over 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Women with signs and symptoms of myocardial ischemia (chest pain, abnormal stress testing, abnormal noninvasive testing) in the absence of obstructive coronary artery disease (epicardial coronary stenosis <50% luminal diameter stenosis).
2. Women with ≥10% myocardial ischemia by CMR perfusion.

Exclusion Criteria:

1. Contraindications to withholding nitrates, beta-blockers, calcium channel agents, ACE/ARB agents for 48 hours prior to testing.
2. Contraindications in CMR including AICD, pacemaker, untreatable claustrophobia or known angio-edema.
3. Contraindications to ranolazine including hepatic insufficiency, prolonged QT, renal failure.
4. Women taking drugs that inhibit CYP3A such as diltiazem, verapamil, ketoconazole, macrolides or HIV protease inhibitors.
5. Women less than 18 years of age.
6. Women on drugs that prolong the QT interval such as Class Ia or III antiarrhythmic agents, erythromycin, certain antipsychotics.
7. Pregnancy or breast feeding.
8. Life expectancy less than 6 months.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noel Bairey-Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- AHSP, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chaitman BR. Ranolazine for the treatment of chronic angina and potential use in other cardiovascular conditions. Circulation. 2006 May 23;113(20):2462-72. doi: 10.1161/CIRCULATIONAHA.105.597500. No abstract available. PMID 16717165
- [Background] Buchthal SD, den Hollander JA, Merz CN, Rogers WJ, Pepine CJ, Reichek N, Sharaf BL, Reis S, Kelsey SF, Pohost GM. Abnormal myocardial phosphorus-31 nuclear magnetic resonance spectroscopy in women with chest pain but normal coronary angiograms. N Engl J Med. 2000 Mar 23;342(12):829-35. doi: 10.1056/NEJM200003233421201. PMID 10727587
- [Background] Doyle M, Fuisz A, Kortright E, Biederman RW, Walsh EG, Martin ET, Tauxe L, Rogers WJ, Merz CN, Pepine C, Sharaf B, Pohost GM. The impact of myocardial flow reserve on the detection of coronary artery disease by perfusion imaging methods: an NHLBI WISE study. J Cardiovasc Magn Reson. 2003 Jul;5(3):475-85. doi: 10.1081/jcmr-120022263. PMID 12882078
- [Background] Hundley WG, Hamilton CA, Thomas MS, Herrington DM, Salido TB, Kitzman DW, Little WC, Link KM. Utility of fast cine magnetic resonance imaging and display for the detection of myocardial ischemia in patients not well suited for second harmonic stress echocardiography. Circulation. 1999 Oct 19;100(16):1697-702. doi: 10.1161/01.cir.100.16.1697. PMID 10525488
- [Background] Hundley WG, Hillis LD, Hamilton CA, Applegate RJ, Herrington DM, Clarke GD, Braden GA, Thomas MS, Lange RA, Peshock RM, Link KM. Assessment of coronary arterial restenosis with phase-contrast magnetic resonance imaging measurements of coronary flow reserve. Circulation. 2000 May 23;101(20):2375-81. doi: 10.1161/01.cir.101.20.2375. PMID 10821813
- [Background] Hundley WG, Morgan TM, Neagle CM, Hamilton CA, Rerkpattanapipat P, Link KM. Magnetic resonance imaging determination of cardiac prognosis. Circulation. 2002 Oct 29;106(18):2328-33. doi: 10.1161/01.cir.0000036017.46437.02. PMID 12403662
- [Background] Johnson BD, Shaw LJ, Buchthal SD, Bairey Merz CN, Kim HW, Scott KN, Doyle M, Olson MB, Pepine CJ, den Hollander J, Sharaf B, Rogers WJ, Mankad S, Forder JR, Kelsey SF, Pohost GM; National Institutes of Health-National Heart, Lung, and Blood Institute. Prognosis in women with myocardial ischemia in the absence of obstructive coronary disease: results from the National Institutes of Health-National Heart, Lung, and Blood Institute-Sponsored Women's Ischemia Syndrome Evaluation (WISE). Circulation. 2004 Jun 22;109(24):2993-9. doi: 10.1161/01.CIR.0000130642.79868.B2. Epub 2004 Jun 14. PMID 15197152
- [Background] Kim RJ, Wu E, Rafael A, Chen EL, Parker MA, Simonetti O, Klocke FJ, Bonow RO, Judd RM. The use of contrast-enhanced magnetic resonance imaging to identify reversible myocardial dysfunction. N Engl J Med. 2000 Nov 16;343(20):1445-53. doi: 10.1056/NEJM200011163432003. PMID 11078769
- [Background] Kim WY, Danias PG, Stuber M, Flamm SD, Plein S, Nagel E, Langerak SE, Weber OM, Pedersen EM, Schmidt M, Botnar RM, Manning WJ. Coronary magnetic resonance angiography for the detection of coronary stenoses. N Engl J Med. 2001 Dec 27;345(26):1863-9. doi: 10.1056/NEJMoa010866. PMID 11756576
- [Background] Nagel E, Lehmkuhl HB, Bocksch W, Klein C, Vogel U, Frantz E, Ellmer A, Dreysse S, Fleck E. Noninvasive diagnosis of ischemia-induced wall motion abnormalities with the use of high-dose dobutamine stress MRI: comparison with dobutamine stress echocardiography. Circulation. 1999 Feb 16;99(6):763-70. doi: 10.1161/01.cir.99.6.763. PMID 9989961
- [Background] Nagel E, Klein C, Paetsch I, Hettwer S, Schnackenburg B, Wegscheider K, Fleck E. Magnetic resonance perfusion measurements for the noninvasive detection of coronary artery disease. Circulation. 2003 Jul 29;108(4):432-7. doi: 10.1161/01.CIR.0000080915.35024.A9. Epub 2003 Jul 14. PMID 12860910
- [Background] Panting JR, Gatehouse PD, Yang GZ, Grothues F, Firmin DN, Collins P, Pennell DJ. Abnormal subendocardial perfusion in cardiac syndrome X detected by cardiovascular magnetic resonance imaging. N Engl J Med. 2002 Jun 20;346(25):1948-53. doi: 10.1056/NEJMoa012369. PMID 12075055
- [Background] Schwitter J, DeMarco T, Kneifel S, von Schulthess GK, Jorg MC, Arheden H, Ruhm S, Stumpe K, Buck A, Parmley WW, Luscher TF, Higgins CB. Magnetic resonance-based assessment of global coronary flow and flow reserve and its relation to left ventricular functional parameters: a comparison with positron emission tomography. Circulation. 2000 Jun 13;101(23):2696-702. doi: 10.1161/01.cir.101.23.2696. PMID 10851206
- [Background] Wahl A, Paetsch I, Gollesch A, Roethemeyer S, Foell D, Gebker R, Langreck H, Klein C, Fleck E, Nagel E. Safety and feasibility of high-dose dobutamine-atropine stress cardiovascular magnetic resonance for diagnosis of myocardial ischaemia: experience in 1000 consecutive cases. Eur Heart J. 2004 Jul;25(14):1230-6. doi: 10.1016/j.ehj.2003.11.018. PMID 15246641
- [Derived] Mehta PK, Goykhman P, Thomson LE, Shufelt C, Wei J, Yang Y, Gill E, Minissian M, Shaw LJ, Slomka PJ, Slivka M, Berman DS, Bairey Merz CN. Ranolazine improves angina in women with evidence of myocardial ischemia but no obstructive coronary artery disease. JACC Cardiovasc Imaging. 2011 May;4(5):514-22. doi: 10.1016/j.jcmg.2011.03.007. PMID 21565740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 subjects were recruited at Cedars-Sinai Medical Center Cardiology outpatient clinic.
Pre-assignment Details: This is a cross-over study. 20 subjects (10 in study drug arm and 10 in placebo arm) completed period 1. In period 2, the 10 subjects who were on study drug in period 1 were on placebo arm in period 2, and the 10 subjects who were on placebo arm in period 1 were on study drug arm in period 2. The 20 subjects had a 2-week wash out in between.
Groups:
- Study Drug Ranexa Then Placebo; Placebo Then Study Drug Ranexa: 20 subjects (10 in study drug arm and 10 in placebo arm) completed period 1. In period 2, the 10 subjects who were on study drug in period 1 were on placebo arm in period 2, and the 10 subjects who were on placebo arm in period 1 were on study drug arm in period 2. The 20 subjects had a 2-week wash out in between.
Period: Period 1
Arm/Group | Study Drug Ranexa Then Placebo | Placebo Then Study Drug Ranexa
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Perod 2
Arm/Group | Study Drug Ranexa Then Placebo | Placebo Then Study Drug Ranexa
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Study drug Ranexa or Placebo.
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 57 [46 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Magnetic Resonance (CMRs)
Description: Cardiac Magnetic Resonance (CMRs) (CMR 1 and CMR 2) end of the 4th week of treatment 1 and treatment 2 respectively, 4 hours after the morning dose of study drug was performed to measure myocardial perfusion defect in percentage.
Time Frame: 4 weeks and 10 weeks
Measure: Median (Full Range); unit: Percentage of ischemic myocardium
Groups:
- Study Drug Ranexa - CMRs (10 CMR 1 and 10 CMR 2); Placebo - CMRs (10 CMR 1 and 10 CMR 2): CMRs (CMR 1 and CMR 2) were performed to test the efficiency of the treatment of the study drug.
Arm/Group | Study Drug Ranexa - CMRs (10 CMR 1 and 10 CMR 2) | Placebo - CMRs (10 CMR 1 and 10 CMR 2)
Number analyzed (Participants) | 20 | 20
Percentage of ischemic myocardium | 11.7 [8.0 to 19.3] | 16.0 [8.6 to 22.7]

2. Secondary Outcome: Seattle Angina Questionnaire (SAQ)
Description: Questionnaires will be completed (SAQ - Seattle Angina Questionnaire) at the end of each treatment period.
  The Seattle Angina Questionnaire (SAQ) is a self-administered, 19-item questionnaire, a cardiac disease-related quality-of-life measure. The SAQ is well validated and sensitive to clinical changes. It has five subscales: physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception. The possible range of scores for each of the five subscales is 0 to 100, with higher scores indicating better quality of life. A change of 10 points in any of the subscales is considered to be clinically important.
  Each final SAQ domain ranges from 0-100, where higher is a better outcome score. Subscales are not combined. Median, SD and range are calculated for each domain.
Time Frame: 4 weeks and 10 weeks
Measure: Median (Full Range); unit: units on a scale
Groups:
- Study Drug: Study drug Ranexa arm
- Placebo: Placebo arm
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Physical Functioning | 91.7 [79.2 to 97.9] | 83.3 [66.6 to 97.2]
  Angina Stability | 75 [50 to 100] | 50 [25 to 75]
  Angina Frequency | 80 [50 to 100] | 75 [60 to 87.5]
  Treatment Satisfaction | 87.5 [75 to 100] | 93.8 [75 to 100]
  Quality of Life | 75 [60.4 to 83.3] | 66.7 [58.3 to 75.0]

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Study Drug | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
This was a pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No